CLINICAL TRIAL: NCT03378102
Title: Antigen Specific Adoptive T Cell Therapy for Refractory Opportunistic Adenovirus Infection After a Hematopoietic Stem Cell Transplantation
Brief Title: Antigen Specific Adoptive T Cell Therapy for Adenovirus Infection After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mari Dallas (Other)
Responsible Party: Sponsor-Investigator, Mari Dallas, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4Z17
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: T Cell Therapy; Opportunistic Infection
MeSH Terms: conditions — Opportunistic Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interferon (IFN)-gamma-secreting HAdV antigen specific T cells (Experimental): Virus-specific, antigen selected cells will be obtained using the CliniMACS® Prodigy System. The donor will be screened for their ability to produce an IFN-gamma- secretion response to HAdV by testing the donor's mononuclear cells with the Miltenyi Rapid Cytokine Inspector kit. Donors with appropriate IFN-gamma secretion response will undergo a steady state leukapheresis. The investigational product (IP) will be generated using the CCS-IFN enrichment program with an approximate duration time of 15 hours. IP will be suspended in 0.9 normal saline + 2.5% albumin and distributed for infusion and infused within 4 hours as a bolus on day 0.
  Subjects will receive virus-specific, antigen selected T cells within a targeted range of 1 x 10^3- 2 x 10^5 per kg of recipient weight.
  Interventions: Biological: IFN-gamma-secreting HAdV antigen specific T cells

INTERVENTIONS:
Biological: IFN-gamma-secreting HAdV antigen specific T cells — Antigen selected cells will be obtained using the CliniMACS(R) Prodigy System from a compatible donor. Isolated cells will be infused into the donor to treat human adenoviral infection after transplant
  Other Names: Antigen-selected, adenovirus-specific T Cells

SUMMARY:
The purpose of this study is to determine if it is possible to treat an infection with a cell-based immunotherapy (therapy that uses the patient's own immune system to treat the infection). This treatment is called adoptive T cell therapy. Another purpose is to learn about the side effects and toxicities of adoptive T cell therapy.

Adoptive T cell therapy is an investigational (experimental) therapy that works by using the blood of a donor that has immunity against the virus. The donor cells are collected and then the cells, called T cells, that are capable of defending against the virus are selected out. These selected T cells are then infused back into the patient, to try to give the immune system the ability to fight the infection. Adoptive T cell therapy is experimental because it is not approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Brief Background/Rationale: This study seeks to determine the feasibility of using antigen specific T cells isolated with the CliniMACS® Cytokine Capture System (CCS) for the treatment of adenovirus infections occurring after allogeneic Hematopoietic Stem Cell Transplantation (HSCT).

Primary Objective: To determine the feasibility of the treatment of opportunistic adenovirus infection after HSCT with adenovirus-specific, antigen-selected T cells, using the CliniMACS® Prodigy System.

Exploratory Objective(s)

* To describe the safety profile of the infusion of virus - specific, antigen selected T cells.
* To describe the toxicities related to infusion of virus - specific, antigen selected T cells.
* To describe the rate of eradication of opportunistic adenovirus infection after treatment with virus-specific, antigen-selected T cells using the CliniMACS® Prodigy System.

Study Design:

This feasibility study will include a single treatment cohort including subjects who have failed to respond, are intolerant or have contraindications to antiviral agents used for treatment of Human Adenovirus (HAdV) (ganciclovir, valganciclovir, foscarnet and cidofovir).

Patients will be enrolled in a staggered pattern to ensure safety.

* Patient 1 will be enrolled and observed for 30 days after infusion of virus specific T cells before enrollment of a subsequent patient.
* Patient 2 will be enrolled ≥ 30 days after treatment of patient 1 and will be observed for 30 days before enrollment of a subsequent patient.
* Subsequent patients will be enrolled in 6 cohorts of 3 subjects each. A safety period between cohorts of 30 days (between treatment of the last subject of one cohort and the first subject of the subsequent cohort).

Study Design: Staggered enrollment of patients with an observation period of 30 days after infusion. Safety monitoring points planned after patient No. 5 and No. 11

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received allogeneic HSCT and be greater than 30 days post-HSCT at the time of registration.
* Patients must have evidence of documented HAdV infection/reactivation. Patients may be:

  * Symptomatic with any detectable viral load OR
  * Asymptomatic with viral load that is:

>1000 copies/ml in peripheral blood OR qualitative detection in stool, urine and/or other specimens

* Patients must have poor response and/or contraindication to therapy:

  * Absence of an improvement of viral load (decrease by at least 1 log, i.e. 10-fold) after ≥ 14 days of antiviral therapy with ganciclovir, valganciclovir and/or foscarnet. OR
  * New, persistent and/or worsening HAdV-related symptoms, signs and/or markers of end organ compromise while on antiviral therapy with ganciclovir, valganciclovir or foscarnet. OR
  * Have contraindications or experience adverse effects of antiviral therapy with ganciclovir, valganciclovir, cidofovir or foscarnet.
* Performance Score: Eastern Cooperative Oncology Group (ECOG) Performance Score ≤ 3. Karnofsky (≥ 16 years) or Lansky (<16 years) performance score ≥ 50
* The effects of virus-specific, antigen-selected T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 4 weeks prior to study entry, for the duration of study participation and for 3 months after completing treatment.
* Subjects who are 14 years and older must have the ability to understand and the willingness to sign a written informed consent document, or assent document.

Exclusion Criteria:

* Pregnant or breastfeeding women are excluded from this study. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with the agents described above, breastfeeding should be discontinued if the mother participates in this trial.
* Patients with opportunistic viral infections other than HAdV.
* Patients with active, grade II-IV, acute graft versus host disease (GVHD), chronic GVHD or any condition requiring high doses of glucocorticosteroid (>0.5 mg/kg/day prednisone or its equivalent) as treatment.
* Treatment with antithymocyte globulin within 28 days of planned infusion of virus - specific, antigen selected T cells.
* Treatment with virus - specific T cells within 6 weeks (42 days) of planned infusion.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with severe adverse events | Up to 100 days after infusion
  This is a measure of feasibility: Severe adverse events are related to the infusion of virus-specific, antigen selected T cells, Grade ≥ 3 acute graft versus host disease,• Death within 30 days of the infusion of the virus-specific, antigen selected T cells that is considered by the investigators to be probably or possibly related to the T cell infusion

SECONDARY OUTCOMES:
Number of patients with viral response | Up to 30 days after infusion
  Clearance: No measurable viral load after therapy Response: Decrease by ≥ 1 log after therapy Persistence: Change by < 1 log after therapy Progression: Increase by ≥1 log after therapy
Number of patients with clinical response | Up to 30 days after infusion
  Clinical Response: Resolution of symptoms and signs of viral infection or reactivation Incomplete clinical response: Improvement, but not resolution of symptoms and signs of viral infection or reactivation Stable clinical disease: No change in symptoms or signs of viral infection Progressive clinical disease: Worsening of symptoms or signs of viral infection
Time from enrollment to T cell product infusion | Up to 24 hours
Time from peripheral mononuclear cell collection to T cell product infusion | Up to 15 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mari H Dallas, MD, Principal Investigator — University Hospitals, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No